CLINICAL TRIAL: NCT01898117
Title: Biomarker Discovery Randomized Phase IIb Trial With Carboplatin-cyclophosphamide Versus Paclitaxel With or Without Atezolizumab as First-line Treatment in Advanced Triple Negative Breast Cancer
Brief Title: Triple-B Study;Carboplatin-cyclophosphamide Versus Paclitaxel With or Without Atezolizumab as First-line Treatment in Advanced Triple Negative Breast Cancer
Acronym: Triple-B
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Borstkanker Onderzoek Groep (Network); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: M13TNB; 2013-001484-23 (EudraCT Number); NL44403.031.13 (Other: CCMO)
Record Dates: First submitted 2013-06-27; First posted 2013-07-12 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Triple negative; Metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Carboplatin; Cyclophosphamide; atezolizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Carbo/cyclo (Active Comparator): Carboplatin AUC=5 Cyclophosphamide 600 mg/m2 Q 4 weeks
  Interventions: Drug: Carbo/cyclo
- Carbo/cyclo + Atezolizumab (Active Comparator): Carboplatin AUC=5 Cyclophosphamide 600 mg/m2 atezolizumab 840 mg d1,15 Q 4 weeks
  Interventions: Drug: Carbo/cyclo + atezolizumab
- Paclitaxel (Active Comparator): Paclitaxel 90 mg/m2 d1, 8, 15 Q 4 weeks
  Interventions: Drug: Paclitaxel
- Paclitaxel + atezolizumab (Active Comparator): Paclitaxel 90 mg/m2 d1, 8, 15 atezolizumab 840 mg d1,15 Q 4 weeks
  Interventions: Drug: Paclitaxel + Atezolizumab

INTERVENTIONS:
Drug: Carbo/cyclo
  Other Names: Carboplatin; Cyclophosphamide
  Arms: Carbo/cyclo
Drug: Carbo/cyclo + atezolizumab
  Other Names: Carboplatin; Cyclophosphamide; Atezolizumab
  Arms: Carbo/cyclo + Atezolizumab
Drug: Paclitaxel
  Arms: Paclitaxel
Drug: Paclitaxel + Atezolizumab
  Other Names: Paclitaxel; Atezolizumab
  Arms: Paclitaxel + atezolizumab

SUMMARY:
Triple negative breast cancer (TNBC) is a difficult to treat molecular subtype with a poor survival. TNBC can be divided into at least two molecular entities; BRCA-like and non-BRCA-like. In this trial we would like to investigate whether a molecular subgroup exists within TNBCs that derives a benefit from atezolizumab added to first line chemotherapy.

DETAILED DESCRIPTION:
Atezolizumab, a humanized monoclonal antibody that targets human programmed death-ligand 1 (PD-L1) has shown activity in TNBC. Early clinical trials with anti-PD-(L)1 monotherapy have shown that the median duration to response in TNBC is remarkably long (18 weeks) compared to cytotoxic chemotherapy. Since advanced TNBC is characterized by rapid disease progression, most patients with TNBC may not have the opportunity to derive benefit from immunotherapy. We hypothesize that by combining atezolizumab with paclitaxel or carboplatin-cyclophosphamide the desired rapid tumor control will be obtained with chemotherapy and subsequently atezolizumab can result in durable responses in a significant subset of patients. It is unknown whether addition of atezolizumab to first line chemotherapy in TNBC is more beneficial than adding this antibody to a second line treatment schedule. Because of this and because of the poor outcome of patients with advanced TNBC experiencing disease progression after first line palliative chemotherapy, patients who were randomized to a chemotherapy only arm in this study will be offered the opportunity to cross over to the other chemotherapy regimen plus atezolizumab at disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Metastasized or locally advanced incurable triple negative breast cancer; patients with stage IV at diagnosis are eligible as well. If the primary lesion is the only measurable lesion according to RECIST criteria, every locoregional treatment must be mentioned to the investigators.
* Histologically confirmed triple negative breast cancer (ER: < 10% nuclear staining of tumor cells on IHC; HER2: either score 0 or 1 at immunohistochemistry or negative at in situ hybridization [CISH or FISH] in case of score 2 or 3 on IHC)
* Histological confirmation of triple negative breast cancer of a metastatic lesion is recommended
* Histological or cytological confirmation of metastatic breast cancer is required in case of normal CA 15.3 levels
* Primary tumor or metastasis tissue (10 x10 μm blank slides FFPE tumor material) sent to NKI-AVL for BRCA-like testing
* Pretreatment histological biopsy of a metastatic lesion for the translational research questions (tumor tissue from bone metastases cannot be used).
* No previous cytotoxic therapy for metastatic disease
* Disease-free interval of at least 12 months after completion of adjuvant paclitaxel or platinum compound therapy
* Disease-free interval of at least 6 months after completion of adjuvant docetaxel
* Measurable disease according to RECIST v1.1
* WHO performance status of 0 or 1
* Adequate bone marrow function: neutrophils ≥ 1.5 x 10E9 cells/l, platelets ≥100 x 10E9 cells/l, Hb ≥ 6.2 mmol/l.
* Normal liver function: bilirubin < 1.5 x upper limit of the normal range (ULN); alkaline phosphatase < 2.5 x ULN (< 5 x ULN in case of liver metastases, and < 7 x ULN in case of bone metastases); transaminases (ASAT/ALAT) < 2.5 x ULN (and < 5 x ULN in case of liver metastases).
* Normal renal function:

  > calculated (Cockcroft-Gault) or measured creatinine clearance > 50 mL/min
* INR < 1.5 and APTT normal, unless patient is on stable anti-coagulant treatment for at least two weeks with a low molecular weight heparin or coumarin, then an INR within the target range (usually between 2 and 3) is allowed.
* Written informed consent

Exclusion Criteria:

* Receptor conversion to hormone receptor positive (defined as >= 10% positive ER or PgR tumor cells) or HER2 positive
* Another cancer except basal-cell carcinoma of the skin or in situ cervical cancer within the previous 5 years
* Other antitumor therapy within the previous 21 days with the exception of endocrine therapy. The patient should have stopped any endocrine therapy before start study treatment.
* Radiotherapy with palliative intent within the previous 7 days before randomization.
* Known CNS disease except for treated brain metastases.
* Uncontrolled serious medical or psychiatric illness
* Pre-existing peripheral neuropathy > grade 1 (NCI-CTC AE (version 4.03)) at inclusion
* Severe infection within 4 weeks prior to randomization
* received antibiotocs within 2 weeks prior to cycle 1, day 1
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to randomization or anticipation of need for major surgical procedure during the course of the study
* New York Heart Association Class II or greater congestive heart failure. LVEF by MUGA, ultrasound or MRI must be ≥ 50% and should be performed within 4 weeks prior to randomization if cardiac failure is suspected.
* History of myocardial infarction or unstable angina within 6 months prior to randomization
* History of myocardial infarction or unstable angina or unstable arrhytmias within 3 months prior to randomization

futher criteria, see protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Validate the BRCA1-like test | assessed up to 120 months
  Validate the BRCA1-like test in predicting differential PFS with first line alkylating and platinum agents (+/- antibody add-on) when compared to paclitaxel (+/- antibody add-on) in TNBC

SECONDARY OUTCOMES:
Determine whether the addition of atezolizumab to paclitaxel is more favorable than adding atezolizumab to carboplatin-cyclophosphamide for patients with PD-L1 positive tumors defined as combined positive score (CPS) 10 or higher (PFS1) | Assessed up to 120 months
  Compare the overal survival (OS), overall response rate (ORR), clinical benefit rate (CBR) and duration of response (DOR) between the groups
Determine whether the addition of atezolizumab to paclitaxel is more favorable than adding atezolizumab to carboplatin-cyclophosphamide (PFS1) | Assessed up to 120 months
  Compare the overal survival (OS), overall response rate (ORR), clinical benefit rate (CBR) and duration of response (DOR) between the groups
Improvement of objective response by adding atezolizumab | assessed up to 120 months
  Determine whether atezolizumab added to first line palliative chemotherapy will result in more objective responses and a higher proportion of patients who are free of progression at 6 months and at 12 months
PD-L1 status (immunohistochemistry) in tumor infiltrating immune cells | Assessed up to 120 months
  Analyze whether PD-L1 status (immunohistochemistry) in tumor infiltrating immune cells predicts for potential differential PFS benefit of atezolizumab added to first line palliative chemotherapy in TNBC
Intratumoral CD8 and/or tumor-infiltrating lymphocytes (TIL) | Assessed up to 120 months
  Analyze whether intratumoral CD8 and/or tumor-infiltrating lymphocytes (TIL) predict for differential PFS benefit of atezolizumab added to first line palliative chemotherapy in TNBC
Compare PFS between alkylating-platinum regimen to paclitaxel as first line chemotherapy in BRCA1-like patients | Assessed up to 120 months
  Evaluate whether an alkylating-platinum regimen is more effective than paclitaxel as first line chemotherapy regarding PFS in BRCA1-like TNBC
Compare PFS between alkylating-platinum regimen to paclitaxel as first line chemotherapy in non BRCA1-like patients | Assessed up to 120 months
  Evaluate whether an alkylating-platinum regimen is more effective than paclitaxel as first line chemotherapy regarding PFS in non BRCA1-like TNBC
TNBC molecular subtypes- based on RNA -expression analysis | Assessed up to 120 months
  define whether different TNBC molecular subtypes- based on RNA -expression analysis - predict for differential PFS benefit of atezolizumab added to first line palliative chemotherapy in TNBC
pretreatment LDH level | Assessed up to 120 months
  define whether pretreatment LDH level predicts for differential benefit of atezolizumab added to first line palliative chemotherapy in TNBC
Define predictive biomarkers for objective response gain | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  Define predictive biomarkers for objective response gain of the addition of atezolizumab to first line chemotherapy; e.g PD-L1, intratumoral CD8, TILs and pre-treatment LDH
Define predictive biomarkers for PFS gain- chemotherapy | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  Define predictive biomarkers for PFS gain of carboplatin-cyclophosphamide or paclitaxel chemotherapy
Define predictive biomarkers for PFS gain - atezolizumab | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  Define predictive biomarkers for PFS gain of addition of atezo lizumab to first line palliative chemotherapy in TNBC
Determine PFS in cross over | At 6 and 12 months and up to 120 months
  Determine the PFS and objective response after cross over to the other chemotherapy regimen with atezolizumab (PFS2)
Overal Response Rate (ORR) | Assessed up to 120 months
  proportion of patients that is free of progression at 6 months and at 12 months after cross-over to the other chemotherapy regimen with atezolizumab
Benefit Atezolizumab | Assessed up to 120 months
  Evaluate whether addition of atezolizumab to chemotherapy in first line is more beneficial than when added in second line
Overall survival (OS) | assessed up to 120 months
  Evaluation of overall survival (OS) for all (sub)group comparisons as pre-specified
Toxicity of all study regimens | Assessed at 1 year
  Adverse events will be graded according to NCI Common Toxicity Criteria version 4.03
Efficay in patients treated with or without Bevacizumab | Assessed up to 120 months
  Evaluate preliminary efficacy by PFS and OS in subgroups of patients treated before amendment 3 with carboplatin/cyclophosphamide or paclitaxel with or without bevacizumab
Determine PFS in BRCA like TNBC | From date of randomization until date of first documented progression or date of death, which ever comes first, assessed up to 120 months
  Determine whether an alkylating platinum regimen is more effective then paclitaxel regarding PFS in BRCA like TNBC
putative predictive potential of BRCA1-like status | Assessed up to 120 months
  Evaluate putative predictive potential of BRCA1-like status in various subgroups defined by treatment regimen received before amendment 3.

CONTACTS AND LOCATIONS:
Overall Officials: Rianne Oosterkamp, MD, Principal Investigator — MC Haaglanden; Marleen Kok, MD, Principal Investigator — NKI-AvL
Locations (49):
- Netherlands (49):
  - MCA, Alkmaar
  - Noordwest Ziekenhuis Groep, Alkmaar
  - ZGT, Almelo
  - Meander Medisch Centrum, Amersfoort
  - BovenIJ, Amsterdam
  - Netherlands Cancer Institute, Amsterdam
  - AZVU, Amsterdam
  - OLVG, Amsterdam
  - Gelre Ziekenhuis, Apeldoorn
  - Rijnstate, Arnhem
  - Lievensberg ziekenhuis, Bergen op Zoom
  - Rode Kruis Ziekenhuis, Beverwijk
  - Amphia, Breda
  - IJsselland ziekenhuis, Capelle aan den IJssel
  - Reinier de Graaf Gasthuis, Delft
  - Deventer ziekenhuis, Deventer
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Nijsmellinghe, Drachten
  - Ziekenhuis Gelderse Vallei, Ede
  - Maxima Medisch Centrum, Eindhoven
  - Catharina ziekenhuis, Eindhoven
  - Jeroen Bosch ziekenhuis, Eindhoven
  - Medisch Spectrum Twente (MST), Enschede
  - Admiraal de Ruyter ziekenhuis, Goes
  - Groene Hart, Gouda
  - Groene Hart Ziekenhuis, Gouda
  - Martini Ziekenhuis, Groningen
  - St. Jansdal, Harderwijk
  - Tergooi ziekenhuizen, Hilversum
  - Spaarne Gasthuis, Hoofddorp
  - Dijklander ziekenhuis, Hoorn
  - MCL, Leeuwarden
  - LUMC, Leiden
  - Haaglanden MC, Leidschendam
  - MUMC, Maastricht
  - St. Antonius ziekenhuis, Nieuwegein
  - Bravis ziekenhuis, Roosendaal
  - St. Fransicus Gasthuis, Rotterdam
  - Ikazia, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
  - Stichting Franciscus Vlietland Groep locatie Gasthuis, Rotterdam
  - Vlietland ziekenhuis, Schiedam
  - Zuyderland, Sittard
  - Haga, The Hague
  - Elisabeth Tweesteden ziekenhuis, Tilburg
  - Diakonessenziekenhuis, Utrecht
  - UMCU, Utrecht
  - VieCuri Medisch Centrum voor Noord-Limburg, Venlo
  - Isala Klinieken, Zwolle

REFERENCES:
- [Derived] Egger SJ, Chan MMK, Luo Q, Wilcken N. Platinum-containing regimens for triple-negative metastatic breast cancer. Cochrane Database Syst Rev. 2020 Oct 21;10(10):CD013750. doi: 10.1002/14651858.CD013750. PMID 33084020